CLINICAL TRIAL: NCT00304382
Title: Humoral Determinants of Immunity to Pneumococcal Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: INDB-013-05F; H-16562 (Other Grant/Funding Number: VA Medical Center, Houston)
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Pneumonia; Pneumococcal Infections; Infections, Streptococcus Pneumoniae
Keywords: Pneumococcus; Pneumococcal pneumonia
MeSH Terms: conditions — Pneumonia; Pneumococcal Infections; Pneumonia, Pneumococcal | interventions — Heptavalent Pneumococcal Conjugate Vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- PPV-PCV (Experimental): Patients receive Pneumovax, and 6 months later Prevnar
  Interventions: Biological: Prevnar; Biological: Pneumovax
- PCV-PPV (Experimental): Patients receive Prevnar, and 6 months later Pneumovax
  Interventions: Biological: Prevnar; Biological: Pneumovax
- PCV-PCV (Experimental): Patients receive Prevnar, and 6 months later Prevnar again
  Interventions: Biological: Prevnar
- PCV only (Experimental): Patients receive Prevnar only
  Interventions: Biological: Prevnar

INTERVENTIONS:
Biological: Prevnar — 0.5 ml IM into each deltoid muscle one time (or two in group PCV-PCV)
  Other Names: Pneumococcal 7-Valent Conjugate Vaccine
Biological: Pneumovax — 0.5 ml IM one time
  Other Names: Pneumococcal Vaccine Polyvalent
  Arms: PCV-PPV; PPV-PCV

SUMMARY:
The purpose of this study is to determine whether there are differences in the level of antibody to capsular polysaccharides of S. pneumoniae or the physiological activity of such antibody after vaccinating patients who have recovered from pneumococcal pneumonia with pneumococcal polysaccharide vaccine (Pneumovax) or conjugate pneumococcal vaccine (Prevnar).

DETAILED DESCRIPTION:
Streptococcus pneumoniae (pneumococcus) is the most common cause of pneumonia leading to hospitalization of adults. Resistance to infection is generally thought to be highly associated with antibody to the capsular polysaccharide (CPS). Most people who develop pneumococcal pneumonia lack antibody to the capsule of the infecting type. We have previously shown that some persons develop this infection despite the presence of antibody to the capsular polysaccharide of the infecting type. When such antibody is found, it tends to be poorly functional (DM Musher et al, J Infect Dis 182:158-167, 2000) in that it opsonizes pneumococci poorly for phagocytosis by human white blood cells in vitro, and protects mice poorly or not at all against challenge with the infecting organism.

About 20% of patients with pneumococcal pneumonia in our previous study had been vaccinated with the only vaccine currently in use for adults, namely 23-valent pneumococcal vaccine (Pneumovax [Merck]). This product consists of purified capsular polysaccharides from 23 different serotypes of S. pneumoniae. During the past two years, with more active vaccination programs at our hospital, the proportion of pneumococcal pneumonia patients who have been vaccinated has increased to about 60%. Clearly, the vaccine has not provided a full degree of protection.

After many years of study, including one involving nearly 40,000 children in the Kaiser Permanent health care system, a new form of pneumococcal vaccine was released. In this vaccine, Prevnar [Wyeth-Lederle], capsular polysaccharide from 7 of the most common pneumococcal types were conjugated to a protein that closely resembles diphtheria toxoid. There have been suggestions that Prevnar stimulates antibody in some subjects who fail to respond to Pneumovax (DM Musher et al, Clin Infect Dis 27:1487-1490, 1998) and also that the resulting antibody may more effectively opsonize bacteria for phagocytosis.

We propose to focus the present research on persons who develop pneumococcal pneumonia, a group that is regarded as being at very high risk of reinfection. Persons who recover from pneumococcal pneumonia will be randomized to vaccination revaccination with Pneumovax or vaccination with Prevnar. These studies will clarify whether administration of protein conjugate pneumococcal vaccine stimulates antibody in patients with pneumonia who failed to respond to prior vaccination or stimulates better functional antibody in those who have previously responded with antibody that is only poorly functional.

Our laboratory and others have shown that Prevnar successfully immunizes adults (Ahmed et al, J Infect Dis 173:83-90, 1996). The vaccine is not officially recommended for adults because antibody levels are the same after Prevnar as after Pneumovax. Such antibody may be more functional; this has not yet been determined. Prevnar contains only 7 antigens whereas Pneumovax contains 23 antigens; thus, it would be less desirable, in general, to administer this vaccine instead of Pneumovax. However, in patients who have developed pneumonia despite having received Pneumovax, the conjugate vaccine may offer an opportunity to stimulate production of effective antibody. In the proposed research, all participants will eventually receive both Pneumovax and Prevnar.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pneumococcal pneumonia
* Age matched controls who have not had pneumococcal pneumonia
* Patients enrolled must be veterans

Exclusion Criteria:

* Patients who do not have the diagnosis of pneumococcal pneumonia based on a clinical syndrome that is consistent with pneumonia and the finding of pneumococcus in blood or sputum or any other sterile site will be excluded
* Women of child-bearing age will be excluded
* Patients who have had a prior reaction to pneumococcal vaccine that they describe as 'severe' will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2006-09-01 (Actual); Study Completion 2012-06-01 (Actual)

PRIMARY OUTCOMES:
Serum will be used to measure antibody to capsular polysaccharide by ELISA and opsonophagocytic activity | 30 days

SECONDARY OUTCOMES:
Serum will be used to measure antibody to capsular polysaccharide by ELISA and opsonophagocytic capacity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Musher, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States